CLINICAL TRIAL: NCT07391215
Title: 5G-PEARL: Paxalisib in Combination With Temozolomide in Patients With High Grade Malignant Brain Tumours Within the 5G Platform
Brief Title: 5G-PEARL: Paxalisib in Malignant Brain Tumours
Acronym: 5G-PEARL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Minderoo Foundation (Unknown); Kazia Therapeutics Limited (Industry); Royal Marsden NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR5814
Record Dates: First submitted 2023-10-05; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Malignant Primary Gliomas; Glioblastoma Multiforme (GBM)
MeSH Terms: conditions — Glioblastoma | interventions — GDC-0084; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1b (Experimental): The Phase 1b will evaluate the safety and tolerability of paxalisib in combination with temozolomide and determine their preliminary antitumour activity in patients with molecularly defined malignant brain tumours.
  Interventions: Drug: Paxalisib; Drug: Temozolomide capsule
- Phase 2 (Experimental): The Phase 2 part of the study will determine the antitumour activity of investigational agents administered at the RP2D in patients with molecularly defined malignant brain tumours.
  Interventions: Drug: Paxalisib; Drug: Temozolomide capsule

INTERVENTIONS:
Drug: Paxalisib — Supplied as 15 mg capsules (35 capsules per bottle).
  Other Names: GDC-0084
Drug: Temozolomide capsule — Temozolomide will be supplied as 5, 20, 100, 140, 180 or 250 mg hard capsules.
  Other Names: Temodal

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and tolerability of paxalisib in combination with temozolomide and to determine the preliminary antitumour activity of the combination therapy. In the Phase 1b of this study parallel biomarker defined arms will be opened in the front-line unmethylated MGMT setting, enrolling 10 patients onto each arm. These patients will be treated with paxalisib in combination with temozolomide (TMZ). The starting dose of paxalisib will be 45mg once a day (OD) with the option of increasing to 60 mg (30 mg BD) in Cycle 2. TMZ will be administered once daily by mouth on days 1 to 5 in a 28-day cycle, with a starting dose of 150mg/m2 during cycles 1 and 2, and subsequent dose escalation to 200mg/m2 at the start of cycle 3 if cycles 1 and 2 have been well tolerated with no significant toxicity.

DETAILED DESCRIPTION:
The clinical trial will be divided into two parts: Phase 1b (proof of concept of hypothesis-driven biomarker-guided therapies) and Phase 2 (preliminary efficacy testing).

This is a study within 5G: A Next Generation AGile Genomically Guided Glioma Modular Platform for proof-of-concept molecular hypothesis testing in patients with high grade malignant brain tumours.

5G-PEARL is a Bayesian multi-centre, multi-arm, open-label, adaptive, seamless Phase 1/2 trial of paxalisib in combination with temozolomide, for patients with malignant brain tumours.

5G-PEARL will recruit patients with glioblastoma (GBM) into two molecularly-defined biomarker arms of patients who have tumours that harbour:

* Hyperactivating PI3K pathogenic mutations in either PIK3CA (p100) or PIK3R1 (p85) as defined by COSMIC.
* PTEN loss as defined by 'two hits' (including either biallelic loss of PTEN, or PTEN LOH + loss of function mutation) NB: Patients with both co-occurring pathogenic PI3K mutation and PTEN loss will be defaulted to the PTEN arm.

Each biomarker arm, within Phase 1, will have robust GO/ADAPT decision points, reviewed by the Safety Review Committee (SRC) to allow for both agility and clear direction for next steps. A 2-stage Bayesian adaptive design will be performed to assess preliminary efficacy.

In the Phase 1b of this study parallel biomarker defined arms will be opened, initially in the front-line unmethylated MGMT setting setting, enrolling 10 patients onto each arm. These patients will be treated with paxalisib in combination with temozolomide. The starting dose of paxalisib will be 45mg once a day (OD) with the option of increasing to 60 mg (30 mg BD) in Cycle 2. TMZ will be administered once daily by mouth on days 1 to 5 in a 28-day cycle, with a starting dose of 150mg/m2 during cycles 1 and 2, and subsequent dose escalation to 200mg/m2 at the start of cycle 3 if cycles 1 and 2 have been well tolerated with no significant toxicity.

Assuming all 'GO' decisions are met, each biomarker arm will recruit a maximum of 32 patients across Phase 1b/2.

ELIGIBILITY:
Inclusion Criteria:

Phase 1b front line mrd cohort:

1. Patients with histologically confirmed advanced WHO Stage IV glioblastoma (per fourth edition 2016). Per the new 2021 fifth edition of WHO Classification of Tumours of the Central Nervous System, this will include:

   • Glioblastoma, IDH-wildtype Grade 4
2. Patients for Phase 1b will need to have consented to the Minderoo Precision Brain Tumour Programme and have whole genome, and transcriptome data available. Patients who have had NHS funded whole genome sequencing and have available frozen tissue stored can be recruited to the study in parallel to consenting to the Minderoo Precision Brain Tumour Programme to have transcriptome analysis done.
3. Patients for the minimal residual disease (mrd) cohort will be eligible following completion of optimal surgery and Stupp based adjuvant chemoradiotherapy as long as they meet all other inclusion/exclusion criteria. Patients will need to commence Cycle 1 Day 1 of the study no later than 6 weeks from the completion of chemoradiotherapy. Patients who are radiologically progressing following chemo-radiotherapy will not be eligible.
4. 16 years or over.
5. Life expectancy of at least 12 weeks.
6. World Health Organisation (WHO) performance status of 0-1.
7. Neurologically stable (eg without a progression of neurological symptoms or requiring escalating doses of systemic steroid therapy within one week prior to cycle 1, day 1.
8. Written (signed or dated) informed consent and be capable of co-operating with treatment and follow up.
9. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week prior to the first dose of either IMP.

   Haemoglobin (Hb): ≥ 9.0 g/dL Absolute neutrophil count: ≥1.5 x 10^9/L Platelet count: ≥100 x 10^9/L Coagulation: INR < 1.5 and APTT <1.5x if not anticoagulated INR stable > 7 days within intended therapeutic range if anticoagulated Bilirubin: ≤1.5 x ULN; participants with Gilbert's syndrome can enrol if conjugated bilirubin is within normal ranges.

   Alanine aminotransferase (ALT) and aspartate aminotransferase (AST): <3 x ULN Albumin: ≥ 28 g/L Creatinine: <1.5 x ULN Sodium: ≥130 mmol/L Potassium, Calcium, Magnesium, phosphate: Within institution normal ranges (replacement is permitted) HbA1C (%): <8.0 Urinary protein: < 1+ on dipstick
10. Female patients with reproductive potential must have a negative serum pregnancy test within 14 days prior to start of trial.
11. Men and women of childbearing potential must agree to comply with the use of a highly effective method of contraception so as to avoid impregnating a partner or becoming pregnant, respectively, during the study, and for at least 180 days after the last dose of either investigational drug. Please, refer to section 4.1 of the Clinical Trials Facilitation and Coordination Group (CTCG) guidance for further details.

Exclusion Criteria:

Phase 1b frontline mrd cohort:

1. Receipt of treatment before the first dose of study drug (Cycle 1 Day 1) within an interval shorter than the following, as applicable:

   * Bevacizumab during the prior 6 weeks
   * Any investigational medicinal product since diagnosis.
   * Tumour treating fields during the prior 6 weeks
2. Prior immune checkpoint inhibitor therapy or vaccine therapy is not permitted. Prior use of any other immune-modulatory investigational agent must be discussed with sponsor team and CI.
3. Ongoing Grade 2 or greater toxicities from pre-existing conditions or from previous treatments.
4. Patients with carcinomatous meningitis, leptomeningeal spread of tumour, spread of tumour to the brain stem or spinal cord.
5. Has evidence of recent intratumoural or peritumoural haemorrhage on baseline MRI. Patients with radiological findings that are stable on at least 2 consecutive MRI scans at least 3 weeks apart will be eligible.
6. History of clinical relevant bleeding disorders, including significant GI bleeding within last 6 months.
7. History of arterial thromboembolism.
8. Recent (within 3 months) deep vein thrombosis or pulmonary embolism or other significant thromboembolism. Venous port of catheter thrombosis or superficial thrombosis are not considered significant. Patients with prior thrombosis (> 3 months ago) on stable anticoagulation are permitted to be enrolled.
9. History of clinically significant cardiac disorders:

   * Myocardial infarction, or New York Heart Association Class II to IV congestive heart failure, within 6 months of the first dose of study drug.
   * Concurrent and clinically significant abnormalities on electrocardiogram (ECG) at Screening, including a corrected QT interval (QTcF >480ms).
10. History of malabsorption syndrome or other conditions that may interfere with enteral absorption. Patients with a history of or active inflammatory bowel disease (eg Crohn's disease or ulcerative colitis). History of gastrointestinal perforation or fistulae.
11. History of uncontrolled diabetes. Patients with controlled diabetes on therapy with HbA1C <8% will be eligible.
12. Has urine protein > 1g/24 hours. Participants with >1+ on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria.
13. Has significant lung disease including pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, active tuberculosis, or history of opportunistic infections (including PCP or CMV pneumonia).
14. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
15. Steroid requirement for neurological symptom control of >3mg Dexamethasone per day (patients will allowed to enrol if they have been on a stable dose of steroids of equivalent or less than 3mg Dexamethasone for at least 5 days prior to Day 1 of Cycle 1).
16. Has received a live vaccine within 30 days of planned start of study therapy. Note: inactive vaccines including COVID vaccines are allowed prior to 1 week of Day 1 of Cycle 1).
17. Current active concurrent malignancy. Cancer survivors who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease recurrence for three years or more and are deemed at negligible risk of recurrence will be eligible.
18. Is a participant or plans to participate on another interventional clinical trial while taking part in this Phase 1 study. Participation in an observational trial would be acceptable.
19. Any other condition which in the investigator's opinion would not make the patient a good candidate for the clinical trial.
20. Exposure to medications (with or without prescriptions), supplements, herbal remedies, or foods with potential for drug-drug interactions with study interventions within 14 days prior to the first dose of study intervention and during the course of therapy, including strong CYP3A4 inhibitors or inducers, due to potential drug-drug interactions with both paxalisib and temozolomide.
21. Major surgery within 4 weeks (excluding placement of vascular access), minor surgery within 2 weeks.
22. Live and attenuated vaccines are not permitted during or within 4 weeks prior to initiation of study treatment.

Inclusion and Exclusion criteria for Phase 2:

1. This will be broadened following an assessment of the safety and tolerability seen in the Phase 1 to be more inclusive and reflective of the real-world population.
2. Patients with any other CNS tumours will only be eligible for defined Phase 2 biomarker arms once a Phase 1b GO decision has been met. Specific eligibility criteria for these tumours will be defined following an amendment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2029-01-19 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1b - Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) in patients with malignant brain tumours | 12 months
  To identify the incidence, nature and severity of adverse events and laboratory abnormalities, with severity determined according to NCI CTCAE v5.0
Phase 1b - To determine the preliminary antitumour activity of the investigational agent administered at the RP2D in patients with molecularly defined malignant brain tumours | 12 months
  Antitumour activity will be defined on the basis of the following outcomes. If any of the following occur, patients will be considered to have clinically benefitted:
  For front line unmethylated GBM (MRD):
  • Progression-free survival (PFS)
Phase 2 - To determine the antitumour activity of investigational agent administered at the RP2D in patients with molecularly defined malignant brain tumours | 24 months
  Antitumour activity will be defined on the basis of the following outcome:
  • Progression-free survival (PFS), defined as the time from enrolment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RANO
Phase 2 - To determine the antitumour activity of investigational agent administered at the RP2D in patients with molecularly defined malignant brain tumours | 24 months
  Antitumour activity will be defined on the basis of the following outcome:
  Overall survival (OS), defined as the time from enrolment to death from any cause

SECONDARY OUTCOMES:
Phase 1b - To identify genetic biomarkers of response in patients with molecularly selected brain tumours | 12 months
  Determine co-occurring genetic biomarkers predicting response.
Phase 2 - To identify genetic biomarkers of response in patients with molecularly selected brain tumours. | 24 months
  Determine co-occurring genetic biomarkers predicting response.
Phase 2 - To assess changes in Quality of Life over time | 12 months
  OS12, defined as the percentage of patients who remained free of death at 12 months from study enrolment
Phase 2 - To assess changes in Quality of Life over time | 6 months
  PFS6, defined as the percentage of patients who remained free of disease progression 6 months from study enrolment
Phase 2 - Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of combination with TMZ when given as standard of care maintenance therapy | 24 months
  To identify the incidence, nature and severity of adverse events and laboratory abnormalities, with severity determined according to NCI CTCAE v5.0
Phase 2 - To assess changes in Quality of Life over time | 24 months
  Global changes over time in health-related quality of life (HRQOL) as assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ C30) (Baseline, end of C1, C3D1).
Phase 2 - To assess changes in Quality of Life over time | 24 months
  Global changes over time in health-related quality of life (HRQOL) as assessed by the 20-item European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Brain Neoplasm module (EORTC QLQ-BN20) (Baseline, end of C1, C3D1)

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Lopez, MD, PhD, Study Director — National Health Service, United Kingdom
Locations (1):
- Royal Marden NHS Foundation Trust, Sutton, United Kingdom